CLINICAL TRIAL: NCT01365182
Title: Improving Urinary Continence and Quality of Life in Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amy Zhang, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASE 14807; 1R01CA127493-01A2 (NIH)
Record Dates: First submitted 2011-05-26; First posted 2011-06-03 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Urinary Incontinence
Keywords: prostate cancer; urinary incontinence; pelvic floor muscle exercise; self-management; behavioral intervention; quality of life
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A biobehavioral interveniton was tested
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BF+SUPPORT (Experimental): a 60-minute session of biofeedback (BF) training in pelvic floor muscle exercises plus 6 biweekly peer support group sessions during 3 months to learn symptom self- management skills
  Interventions: Behavioral: BF+SUPPORT
- BF+PHONE (Experimental): a 60-minute session of biofeedback (BF) training in pelvic floor muscle exercises plus 6 biweekly individual telephone contact with a therapist during 3 months to learn symptom self- management skills
  Interventions: Behavioral: BF+PHONE
- Usual Care (No Intervention): Subjects continued receiving usual care without receiving any intervention training sessions

INTERVENTIONS:
Behavioral: BF+SUPPORT — A session of biofeedback-assisted pelvic floor muscle exercises (PFME) plus 6 group sessions of the Problem-Solving Therapy (teaching self-management skills).
  Arms: BF+SUPPORT
Behavioral: BF+PHONE — A session of biofeedback-assisted pelvic floor muscle exercises (PFME) plus 6 telephone sessions of the Problem-Solving Therapy (teaching self-management skills).
  Arms: BF+PHONE

SUMMARY:
This intervention program combines biofeedback PFME with a telephone or support group intervention to treat persistent urinary incontinence (UI). The study's primary aims are to improve continence, quality of life, and mood through enhancing adherence to PFME and self-management of incontinence symptoms. The secondary aims are to examine the physiological effects and cost effectiveness of the proposed interventions.

DETAILED DESCRIPTION:
This is a randomized, controlled longitudinal study. Patients with early-stage prostate cancer and UI for more than six months were randomly assigned to one of three study arms: (1) biofeedback PFME plus a support group (BF+SUPPORT); (2) biofeedback PFME plus telephone (BF+PHONE); and (3) usual care (UC). The BF+SUPPORT and BF+PHONE participants learned PFME through computerized biofeedback. Thereafter, the BF+SUPPORT participants attended six group meetings and the BF+PHONE participants had six phone contacts every other week for three months. The UC participants did not receive biofeedback PFME or telephone/group intervention but continued receiving usual medical care. All subjects were assessed blind at baseline, 3 months (post intervention) and 6 months (follow-up). In addition, 49 moderately to severely incontinent patients were recruited from the three study groups to undergo urodynamic testing at baseline and 3 months for the evaluation of physiological changes. Data of the costs for the interventions and the participants' medical care were collected for a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with early stage (I-III) prostate cancer.
2. Have completed cancer treatments six months prior.
3. Presence of incontinence symptoms

Exclusion Criteria:

1. Receiving hormonal treatment.
2. Urinary tract infection or urinary retention.
3. Cognitive impairment.
4. Having an implant

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zhang, Ph.D., Principal Investigator — Case Western Reserve University

REFERENCES:
- [Background] Balch CM, Gershenwald JE, Soong SJ, Thompson JF, Atkins MB, Byrd DR, Buzaid AC, Cochran AJ, Coit DG, Ding S, Eggermont AM, Flaherty KT, Gimotty PA, Kirkwood JM, McMasters KM, Mihm MC Jr, Morton DL, Ross MI, Sober AJ, Sondak VK. Final version of 2009 AJCC melanoma staging and classification. J Clin Oncol. 2009 Dec 20;27(36):6199-206. doi: 10.1200/JCO.2009.23.4799. Epub 2009 Nov 16. PMID 19917835
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Zhang AY, Bodner DR, Fu AZ, Gunzler DD, Klein E, Kresevic D, Moore S, Ponsky L, Purdum M, Strauss G, Zhu H. Effects of Patient Centered Interventions on Persistent Urinary Incontinence after Prostate Cancer Treatment: A Randomized, Controlled Trial. J Urol. 2015 Dec;194(6):1675-81. doi: 10.1016/j.juro.2015.07.090. Epub 2015 Jul 29. PMID 26231554
- [Result] Zhang AY, Fu AZ, Moore S, Zhu H, Strauss G, Kresevic D, Klein E, Ponsky L, Bodner DR. Is a behavioral treatment for urinary incontinence beneficial to prostate cancer survivors as a follow-up care? J Cancer Surviv. 2017 Feb;11(1):24-31. doi: 10.1007/s11764-016-0557-0. Epub 2016 Jun 24. PMID 27341843
- [Result] Zhang AY, Ganocy S, Fu AZ, Kresevic D, Ponsky L, Strauss G, Bodner DR, Zhu H. Mood outcomes of a behavioral treatment for urinary incontinence in prostate cancer survivors. Support Care Cancer. 2019 Dec;27(12):4461-4467. doi: 10.1007/s00520-019-04745-w. Epub 2019 Mar 22. PMID 30903368
- [Result] Zhang AY, Burant C, Fu AZ, Strauss G, Bodner DR, Ponsky L. Psychosocial mechanisms of a behavioral treatment for urinary incontinence of prostate cancer survivors. J Psychosoc Oncol. 2020 Mar-Apr;38(2):210-227. doi: 10.1080/07347332.2019.1678547. Epub 2019 Nov 24. PMID 31762400
- [Result] Zhang AY, Fu AZ. Cost-effectiveness of a behavioral intervention for persistent urinary incontinence in prostate cancer patients. Psychooncology. 2016 Apr;25(4):421-7. doi: 10.1002/pon.3849. Epub 2015 May 12. PMID 25963381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, controlled, longitudinal clinical trial was performed from 2010 to 2013 in Cleveland, Ohio
Groups:
- BE+Support: a 60-minute session of biofeedback (BF) training in pelvic floor muscle exercises plus 6 biweekly peer support group sessions during 3 months to learn symptom self- management skills
Period: Overall Study
Arm/Group | BE+Support | BF+PHONE | Usual Care
Started | 91 | 94 | 94
Completed | 81 | 81 | 82
Not Completed | 10 | 13 | 12
Not completed — Withdrawal by Subject | 10 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BF+Support | BF+PHONE | Usual Care | Total
Number analyzed (Participants) | 81 | 81 | 82 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is measured in years
  years | 66.8 (7.2) | 64.3 (7.3) | 64.9 (8.2) | 65 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Self reported and verified with medical chart data Population: Each row represents a study arm/ group. Total participants from three study arms =244 (overall number of participants)
  Participants
    Gender: Female | 0 | 0 | 0 | 0
    Gender: Male | 81 | 81 | 82 | 244
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: row 1 = overall (n=244) row 2-3: each row represents a study arm/ group
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Race: Asian | 0 | 1 | 1 | 2
    Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Race: Black or African American | 31 | 26 | 28 | 85
    Race: White | 49 | 53 | 51 | 153
    Race: More than one race | 0 | 0 | 0 | 0
    Race: Unknown or Not Reported | 1 | 1 | 2 | 4
Marriat Status (Married) [Count of Participants; unit: Participants] | 54 | 52 | 52 | 158
Education [Count of Participants; unit: Participants]
  Colleage or higher | 27 | 35 | 28 | 90
  High school, associate degree | 46 | 39 | 47 | 132
  Less than high school | 8 | 7 | 7 | 22
Employed [Count of Participants; unit: Participants] | 28 | 43 | 36 | 107
Cancer Stage [Count of Participants; unit: Participants] — The cancer stages were obtained from chart reviews. The stages were determined by treating physicians using the AJCC (American Joint Committee on Cancer) TNM staging system. Stage ranges from 1 to 4, with 4 indicating metastasis (worst) stage. Stage 4 was excluded from this study based on eligibility criteria.
  Participants
    Participants at stage I or II | 77 | 76 | 78 | 231
    Participants at stage III | 4 | 5 | 4 | 13
Received Surgery [Count of Participants; unit: Participants] | 43 | 43 | 47 | 133
Received Radiation [Count of Participants; unit: Participants] | 45 | 43 | 39 | 127
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index "BMI" was collected from medical chart review. "BMI" is typically presented with Unit of Measure "kg/m^2" If your BMI is less than 18.5, it falls within the underweight range. If your BMI is 18.5 to <25, it falls within the healthy weight range. If your BMI is 25.0 to <30, it falls within the overweight range. If your BMI is 30.0 or higher, it falls within the obesity range.
  kg/m^2 | 28.3 (4) | 29.3 (5.7) | 29.2 (5.4) | 28.8 (5)
PSA [Mean (Standard Deviation); unit: ng/mL] — Prostate-specific antigen "PSA" is typically presented with Unit of Measure ng/mL.
  At NIH website, https://www.cancer.gov/types/prostate/psa-fact-sheet, it says "PSA is a protein produced by normal, as well as malignant, cells of the prostate gland. This test measures the level of PSA in the blood," with a higher level indicating a potential problem.
  ng/mL | 0.74 (1.9) | 0.71 (1.7) | 0.49 (1.3) | 0.71 (1.8)
Charlson comorbidity index score [Mean (Standard Deviation); unit: score on a scale] — The Charlson Comorbidity Index (CCI) is a checklist that comprised of 19 health conditions (dichotomously coded as "yes/ no"). The CCI score is a calculated score that assigns different weights to each possible comorbid condition (e.g., myocardial infarction scoring 1, metastatic solid tumor scoring 6). The 19 health conditions were obtained from medical chart reviews. Range of CCI adjusted for age is 0 to 37. Higher CCI scores represent more comorbid conditions and worse projected health outcomes.
  score on a scale | 0.63 (1.1) | 0.78 (1.1) | 0.95 (1.8) | 0.78 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Urinary Leakage
Description: Amount of leakage measured on 1-hour pad test
Time Frame: Measured at baseline, 3 months after baseline, and then 6 months after the baseline assessment
Population: Data are reported only for those who completed the entire study.
Measure: Mean (Standard Deviation); unit: grams
Groups:
- BF+Telephone: a 60-minute session of biofeedback (BF) training in pelvic floor muscle exercises plus 6 biweekly individual telephone contact with a therapist during 3 months to learn symptom self- management skills
Arm/Group | Usual Care | BF+Telephone | BF+Support
Number analyzed (Participants) | 70 | 62 | 67
grams
  T1 (baseline) | 23.2 (48.4) | 22.3 (47.6) | 31.5 (62.9)
  T2 (3 month) | 11 (24.2) | 23.2 (73.5) | 17.9 (43.3)
  T3 (6 month) | 14.2 (37.1) | 7.5 (21.8) | 14.9 (40.1)

2. Primary Outcome: Frequency of Daily Urinary Leakage
Description: Average times of daily leakage measured on a 3-day diary
Time Frame: Measured at baseline, 3 months after baseline, and then 6 months after the baseline assessment
Population: Data are reported only for those who completed this measure at all three assessment points. Subjects that did not complete this measure three times were not included.
Measure: Mean (Standard Deviation); unit: Leaks per day
Groups:
- Usual Care: A control group
- BF+Telephone: Biofeedback plus biweekly telephone (dyad) meeting
- BF+Support: Biofeedback plus biweekly support group meeting
Arm/Group | Usual Care | BF+Telephone | BF+Support
Number analyzed (Participants) | 55 | 49 | 54
Leaks per day
  T1 (baseline) | 3.2 (3.4) | 2.9 (3.0) | 2.7 (3.4)
  T2 (3 month) | 2.8 (3.4) | 1.8 (2.5) | 1.7 (2.7)
  T3 (6 month) | 2.5 (3.0) | 1.7 (2.7) | 1.9 (3.3)

ADVERSE EVENTS:
Time Frame: 7 months (study duration)
Description: This is a behavioral study and has a low risk for study subjects. All participants' charts are reviewed and adverse events are reported.
Arm/Group | BF+Support | BF+PHONE | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/81 | 2/81 | 1/82
Other Adverse Events (participants affected / at risk) | 0/81 | 0/81 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF+Support (N=81) | BF+PHONE (N=81) | Usual Care (N=82)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) — Two urinary tract infection possibly associated with study procedure
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0) — Patient fell during 1-hour pad testing that requires walking for a few minutes.

LIMITATIONS AND CAVEATS:
Limitations:

* The rate of missing data at 6 months was higher for daily leakage frequency than the leakage amount.
* The 3-month intervention duration limited our ability to assess intervention sustainability and long-term effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2009-12-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT01365182/ICF_000.pdf